CLINICAL TRIAL: NCT02062073
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of Abametapir Lotion in Healthy Volunteers Using a Repeat Insult Patch Test Design
Brief Title: Dermal Safety Study to Evaluate the Sensitizing Potential of Abametapir Lotion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: TKL Research, Inc. (Industry); Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ha03-006
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Head Lice
Keywords: head lice; Hatchtech
MeSH Terms: interventions — Sodium Dodecyl Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Abametapir Lotion 0.74% (Active Comparator): 0.2 mL applied topically to the infrascapular area of the back under occlusive patch conditions 3 times weekly for 3 weeks, following with rest period and a challenge.
  Interventions: Drug: Abametapir Lotion 0.74% w/w
- Vehicle Lotion (Placebo Comparator): 0.2 mL applied topically to the infrascapular area of the back under occlusive patch conditions 3 times weekly for 3 weeks, following with rest period and a challenge.
  Interventions: Other: Vehicle Lotion
- 0.1% sodium lauryl sulfate (Other): Concurrent control 0.2 mL applied topically to the infrascapular area of the back under occlusive patch conditions 3 times weekly for 3 weeks, following with rest period and a challenge.
  Interventions: Other: 0.1% sodium lauryl sulfate
- Saline 0.9% (Other): Concurrent control 0.2 mL applied topically to the infrascapular area of the back under occlusive patch conditions 3 times weekly for 3 weeks, following with rest period and a challenge.
  Interventions: Other: saline 0.9%

INTERVENTIONS:
Drug: Abametapir Lotion 0.74% w/w
  Arms: Abametapir Lotion 0.74%
Other: 0.1% sodium lauryl sulfate
  Arms: 0.1% sodium lauryl sulfate
Other: saline 0.9%
  Arms: Saline 0.9%
Other: Vehicle Lotion
  Arms: Vehicle Lotion

SUMMARY:
Purpose of this study will be to determine the potential of abametapir lotion to induce sensitization by repeated topical application to the healthy skin of humans under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Are healthy (to be confirmed by medical history) males or females, 18 years of age or older;
2. In the case of females of childbearing potential, are using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy). Abstinence or vasectomized partner are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
3. If female of childbearing potential, have a negative urine pregnancy test at Day 1, and are willing to submit to a pregnancy test at the end of study;
4. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events;
5. Are of any skin type or race, providing the skin pigmentation will allow discernment of erythema;
6. Complete a patch study Medical Screening form as well as a Medical Personal History form; and
7. Read, understand, and provide signed informed consent.

Exclusion Criteria:

1. Have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction;
2. Are not willing to refrain from using topical/systemic analgesics such as aspirin (daily use of 81 mg aspirin is acceptable), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
3. Are using inhaled/systemic/topical corticosteroids in the 3 weeks prior to and during the study, or systemic/topical antihistamines for 72 hours prior to and during the study;
4. Are using medication which, in the opinion of the investigative personnel, will interfere with the study results, including anti-inflammatory medications;
5. Are unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions, or similar products on the back during the study;
6. Have psoriasis and/or active atopic dermatitis/eczema;
7. Are females who are pregnant, plan to become pregnant during the study, or are breast-feeding a child;
8. Have a known sensitivity to constituents present in the material being evaluated;
9. Have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
10. Have received treatment for any type of internal cancer within 5 years prior to study entry;
11. Have a history of, or are currently being treated for skin cancer;
12. Are currently participating in any other clinical trial;
13. Have any known sensitivity to adhesives; and/or
14. Have received any investigational treatment(s) within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
to evaluate the sensitizing potential of abametapir lotion using repeat insult patch test design | 8 weeks
  Evaluation of dermal reactions at the application sites will be assessed clinically using a visual scale that rates the degree of erythema, edema, and other signs of cutaneous irritation

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dosik, Principal Investigator — TKL Research
Locations (1):
- TKL Reserach, Paramus, New Jersey, United States